CLINICAL TRIAL: NCT04656964
Title: The Safety and Effectiveness of Remimazolam Tosilate Versus Midazolam in Elderly Patients Undergoing Gastrointestinal Endoscopy: A Multicenter ,Prospective, Double-Blinded, Randomized Controlled Study
Brief Title: Comparison Between Remimazolam Tosilate and Midazolam in Elderly Patients Undergoing Gastrointestinal Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Emergency General Hospital (Other); Fenyang Hospital Affiliated to Shanxi Medical University (Unknown)
Responsible Party: Principal Investigator, Yi Feng, MD, Chief of Anesthesiology department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020PHB249-01
Record Dates: First submitted 2020-11-05; First posted 2020-12-07 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Elderly Patients; Gastrointestinal Endoscopy; Midazolam; Remimazolam
Keywords: Remimazolam tosilate; Midazolam; postsedation effect; postsedation safety; cognition function; patients' satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Tosilate group (Experimental): Patients received remimazolam tosilate to maintain sufficient sedation (sufficient sedation as judged by MOAA/S ≤ 4 for 3 consecutive measurements) during endoscopy procedure. And patients were slowly injected of 0.4 ug/kg of remifentanil for 1 min during the examination.When the analgesia was insufficient, Remifentanil can be added 5-10 ug each time according to the situation.
  Interventions: Drug: remimazolam tosilate group
- Midazolam group (Active Comparator): Patients received midazolam to maintain sufficient sedation (sufficient sedation as judged by MOAA/S ≤ 4 for 3 consecutive measurements) during endoscopy procedure. And patients were slowly injected of 0.4 ug/kg of remifentanil for 1 min during the examination.When the analgesia was insufficient, Remifentanil can be added 5-10 ug each time according to the situation.
  Interventions: Drug: Midazolam group

INTERVENTIONS:
Drug: remimazolam tosilate group — Patients received an initial dose of 0.2mg/kg of remimazolam tosilate(plus repeated 2.5 mg top-ups doses to a total of up to 12.5mg within 15 minutes).
  Arms: Remimazolam Tosilate group
Drug: Midazolam group — Patients received an initial dose of 0.03mg/kg of midazolam(One additional dose of 0.015 mg / kg midazolam was allowed).
  Arms: Midazolam group

SUMMARY:
Midazolam is a commonly used drug in gastrointestinal endoscopy due to the good cardiovascular stability and mild respiratory depression for elderly patients. However, there is the concern about the the longer and less predictable recovery or the potential for repeat sedation when the active metabolite becomes bioavailable. Remimazolam Tosilate is an innovative benzodiazepine with better sedation effect and less recovery or resedation issues than midazolam, which possibly make the drug more suitable in elderly patients. We aim to clarify whether remimazolam tosilate is better than midazolam in elderly patients undergoing gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Before starting the endoscopy procedures, patients were randomized to receive remimazolam tosilate or midazolam to maintain sufficient sedation, then remifentanil was slowly injected for patients' sufficient analgesia during the examination. We aim to use patients' recovery time, cognition function and other measurement scales to clarify whether remimazolam tosilate is better than midazolam in elderly patients undergoing gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to undergo a routine diagnostic or therapeutic gastrointestinal endoscopy ;
2. Age 60 to 75 ;
3. ASA physical status score of I, II or III;
4. A body mass index (BMI) of 19 to 28 kg/m2;
5. Systolic blood pressure of 90-140mmHg, diastolic blood pressure of 50-90mmHg, resting heart rate of 50-100bpm and blood pulse oxygen saturation ≥95%

Exclusion Criteria:

1. Those who are refused to be included;
2. Those who are allergic to the drugs used in this study;
3. Epilepsy and other mental illnesses, a history of addiction such as opiates and other analgesics and/or tranquilizers (hypnotics);
4. Severe cardiac dysfunction: NYHA cardiac functions grade 3-4, a history of recent myocardial infarction or cerebral infarction, severe conduction block or malignant arrhythmia;
5. Renal failure or liver cirrhosis;
6. Severe lung infection or upper respiratory tract infection;
7. Sleep apnea syndrome, difficult airway (Mallampati score of 3 or 4) or asthma status;
8. Advanced cancer accompanied by extensive intra-abdominal metastasis, acute and chronic obstruction of the gastrointestinal tract, bleeding and severe abdominal effusion;

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Recovery time after operation | Day 0
  First of 3 consecutive MOAA/S scores of 5 after the last injection of study drug.

SECONDARY OUTCOMES:
Supine heart rate[HR] | Day 0
  Supine heart rate[HR] in (times)
Modified Observer's Assessment of Alertness/Sedation[MOAA/S] | Day 0
  MOAA/S score ranges from 0 to 5 points, 0 point means patients do not respond to noxious stimulation; 5 point means patients responds readily to name spoken in normal tone. When the Modified Observer's Assessment of Alertness/Sedation [MOAA/S] ≤4 that patients are sufficiently sedated.
Visual analogue scale (VAS) | Day 0
  The visual analogue scale (VAS) score ranges from 0 to 10 points (0mm means patients feel no pain, 100mm means patients feel the most severe pain imaginable)
Post-anesthesia discharge score (PADS) | Record within 2 hours ，no more than 6 hours
  Post-anesthesia discharge score PADS score ranges from 0 to 10 points. only when the PADS score≥9 that will the patients leave the post-anesthesia care unit(PACU).
Perioperative anesthesia effect | Day 0
  Induction time（from the drug administration to the start of endoscopy insertion); procedure time(from the endoscopy insertion to the end of procedure);PACU last time(from the entry to PACU to the PADS score≥9).
Drug dosages | Day 0
  The total single dosage of midazolam, propofol, remifentanil and remimazolam tosilate.
Simple Intelligence Assessment Scale (mini-cog) | Every 4 hours, up to 1 week.
  1. Ask the subjects to listen carefully and memorize 3 unrelated words, and then repeat (Apple, Watch, Coin);
  2. Ask the subjects to draw the shape of the clock on a blank sheet of paper, and give the subject a time to mark it on the clock (the CDT of the clock drawing test is correct; it can correctly indicate the sequence of the digits and display the given Fixed time);
  3. Ask the subject to say the 3 words given previously.
Patient overall satisfaction and surgeon satisfaction score | Day 0
  The patient's overall satisfaction score and surgeon satisfaction score were evaluated by 1-10 points (1mm=completely dissatisfied, 100mm=completely satisfied).
Systolic, diastolic, and mean blood pressure [MBP] | Day 0
  Systolic, diastolic, and mean blood pressure [MBP] in(mmHg)
Assessment of pulse oximetry measurements[SpO2] | Day 0
  Assessment of pulse oximetry measurements[SpO2]in(%)
Respiration rate[RR] | Day 0
  Respiration rate[RR] in (times)
End-tidal carbon dioxide [EtCO2] | Day 0
  End-tidal carbon dioxide [EtCO2] in (%)
Rate of coughing and vomiting | Within 24 hours
  Rate of coughing and vomiting in（%）
Level of hypoxia | Within 24 hours
  Oxygen saturation <90% for more than 1 minute ，that share a common Unit of Measure in（%）
Respiratory depression | Within 24 hours
  Respiratory rate < 8 breaths per minute ,that share a common Unit of Measure in（times）
Abdominal pain and nausea | Within 24 hours
  Abdominal pain and nausea in （%）

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China